CLINICAL TRIAL: NCT01259505
Title: Phase I Study of Multiple-Vaccine Therapy Using Epitope Peptides Restricted to HLA-A*2402 in Treating Patients With Refractory Breast Cancer
Brief Title: Safety Study of Multiple-Vaccine to Treat Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tokyo Medical University (Other)
Collaborators: Tokyo University (Other); Saint Luca International Hospital (Unknown)
Responsible Party: Principal Investigator, Minoru Fujimori, Professor, Tokyo Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBCCTA-001-STT
Record Dates: First submitted 2010-12-11; First posted 2010-12-14 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Metastatic Breast Cancer
Keywords: no number
MeSH Terms: conditions — Breast Neoplasms | interventions — KIF20B protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Safety (Experimental): CDCA1，URLC10，KIF20A，DEPDC1 and MPHOSPH1 peptides mixed with Montanide ISA 51 Patients will be vaccinated once a week until patients develop progressive disease or unacceptable toxicity. On each vaccination day, CDCA1，URLC10，KIF20A，DEPDC1 and MPHOSPH1 peptides (0.5, 1 or 2mg of each peptide) mixed with Montanide ISA 51 will be administered by subcutaneous injection.
  Interventions: Biological: CDCA1，URLC10，KIF20A，DEPDC1 and MPHOSPH1

INTERVENTIONS:
Biological: CDCA1，URLC10，KIF20A，DEPDC1 and MPHOSPH1 — CDCA1，URLC10，KIF20A，DEPDC1 and MPHOSPH1 peptides mixed with Montanide ISA 51 Patients will be vaccinated once a week until patients develop progressive disease or unacceptable toxicity. On each vaccination day, CDCA1，URLC10，KIF20A，DEPDC1 and MPHOSPH1 peptides (0.5, 1 or 2mg of each peptide) mixed with Montanide ISA 51 will be administered by subcutaneous injection.

SUMMARY:
The purpose of this study is to evaluate the safety of HLA-A*2402 restricted epitope peptides CDCA1，URLC10，KIF20A，DEPDC1 and MPHOSPH1 emulsified with Montanide ISA 51.

DETAILED DESCRIPTION:
CDCA1，URLC10，KIF20A，DEPDC1 and MPHOSPH1 have been identified as cancer specific molecules especially in breast cancer using genome-wide expression profile analysis by cDNA microarray technique. We have determined the HLA-A*2402 restricted epitope peptides derived from these molecules and identified that these peptides significantly induce the effective tumor specific CTL response in vitro and vivo. According to these findings, in this trial, we evaluate the safety, immunological and clinical response of these peptides. Patients will be vaccinated once a week until patients develop progressive disease or unacceptable toxicity. On each vaccination day, CDCA1，URLC10，KIF20A，DEPDC1 and MPHOSPH1 peptides (0.5, 1 or 2mg of each peptide) mixed with Montanide ISA 51 will be administered by subcutaneous injection. Repeated cycles of vaccine will be administered until patients develop progressive disease or unacceptable toxicity, whichever occurs first. In the phase I study, we evaluate the safety and tolerability of these peptides vaccine. Also we evaluate the immunological and clinical response of this vaccine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or recurrent breast cancer
* Resistant against anthracycline-based and taxane-based chemotherapy or difficult to continue the chemotherapy due to intolerable side effect(s)
* Resistant against trastuzumab or difficult to continue it due to intolerable side effect(s) when her-2 is positive
* ECOG performance status 0-2
* Life expectancy > 3 months
* HLA-A*2402
* Laboratory values as follows

  * 2000/mm3<WBC<15000/mm3
  * Platelet count>100000/mm3
  * Bilirubin < 3.0mg/dl
  * Asparate transaminase < 150IU/L
  * Alanine transaminase < 150IU/L
  * Creatinine < 3.0mg/dl
* Able and willing to give valid written informed consent

Exclusion Criteria:

* Pregnancy(woman of childbearing potential:Refusal or inability to use effective means of contraception)
* Breastfeeding
* Active or uncontrolled infection
* Concurrent treatment with steroids or immunosuppressing agent
* Prior chemotherapy,radiation therapy, or immunotherapy within 4 weeks
* Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-12; Primary Completion 2012-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
safety (Phase I: toxicities as assessed by NCI CTCAE version3) | 1 month

SECONDARY OUTCOMES:
to evaluate efficacy (feasibility as evaluated by RECIST) | 2 months
  to evaluate overall survival to evaluate progression free survivial to evaluate efficacy (feasibility as evaluated by RECIST) to evaluate immunological responses to evaluate quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo Medical University Ibaraki Medical Center, Ami Inashiki, Ibaraki, Japan